CLINICAL TRIAL: NCT02879526
Title: Chidamide Combined With Cyclophosphamide, Prednisone, Thalidomide in Treatment of Fragile Patients With Relapse/Refratory Peripheral T Cell Lymphoma :a Phase II, Single-arm, Open-label, Muti-center Study
Brief Title: Chidamide Combined With Cyclophosphamide, Prednisone, Thalidomide in Treatment of Fragile Patients With Relapse/Refratory Peripheral T Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, WEI XU, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JSPH-003
Record Dates: First submitted 2016-08-21; First posted 2016-08-25 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Relapse/Refratory Peripheral T Cell Lymphoma
Keywords: Relapse/Refratory Peripheral T Cell Lymphoma; Chidamide; Cyclophosphamide、Prednisone、Thalidomide(CPT)
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- C-CPT (Experimental)
  Interventions: Drug: C-CPT

INTERVENTIONS:
Drug: C-CPT — Chidamide 30mg ，twice a week Prednisone 20mg qd Cyclophosphamide 50mg qd Thalidomide 100mg qd

SUMMARY:
The purpose of this study is to investigate efficacy and safety of Chidamide Combined With Cyclophosphamide,Prednisone,Thalidomide in Treatment of Fragile Patients With Relapse/Refratory Peripheral T Cell Lymphoma :a Phase II,Single-arm,Open-label, Muti-center Study

DETAILED DESCRIPTION:
Chidamide is a new histone deacetylase inhibitor and shows anti-tumor activity in Relapse/Refratory Peripheral T Cell Lymphoma.Cyclophosphamide,Prednisone,Thalidomide(CPT) is an oral combination regimen for lymphoma patients who can not stand the standard chemotherapy. The investigators therefore design this open-label,phase II, single-arm trial to investigate the efficacy of Chidamide Combined With CPT in treatment of fragile Patients With Relapse/Refratory Peripheral T Cell Lymphoma

Primary Outcome Measures:

• overall response rate

Secondary Outcome Measures:

* duration of response
* progression free survival
* overall survival Enrollment:45 Study Start Date: August 2016 Primary Completion Date: March 2018

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed Peripheral T Cell Lymphoma,exclude NK/T cell lymphoma
2. Relapse or refractory to at least one prior therapy(chemotherapy or stem cell transplantation)
3. can not
4. age between 18 and 75, both gender
5. ECOG PS 0-1
6. Peripheral ANC >1.5*109/L; platelet >70*109/L; Hb≥ 90g/L
7. Anticipated survival ≥ 3 months
8. No chemotherapy ,radiotherapy and stem cell transplantation within 4 weeks before inclusion
9. Sign in informed consent form, adherence to the study visit schedule and other protocol requirements

Exclusion Criteria:

1. Pregnant women or women in suckling period or with Potentia Generand but not willing to take contraceptives
2. New York Heart Association class III or IV cardiac failure; or history of following disease in past 6 months: acute coronary syndrome, acute heart failure, severe ventricular arrhythmia
3. Poor hepatic function, defined as total bilirubin more than 1.5 fold of upper normal level, ALT, AST more than 2 fold of upper normal level or more than 5fold of upper normal level with hepatic involvement;Poor renal function, defined as serum creatinine more than 1.5 fold of upper normal level
4. CNS or meningeal involvement
5. intervention on myelosuppression within7 days before inclusion
6. patients with active bleeding
7. Major surgery within three weeks before inclusion
8. Positive HIV, syphilis,HCV, or HBV virus load(HBV DNA)> 1×105 copies/ml;
9. Any psychological conditions which may disturb consent.
10. In any conditions which investigator considered ineligible
11. Known sensitivity or allergy to investigational Product.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-06 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | One-year
  overall response rate after treated by C-CPT

SECONDARY OUTCOMES:
Duration of response | One-year
  from the date of response to date of progression, relapse,
Progress-free survival | One-year
  from date of inclusion to date of progression, relapse, or death from any cause
Overall survival | One-year
  from the date of inclusion to date of death, irrespective of cause

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xu, M.D., Ph.D., Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (2):
- China (2):
  - HuaiAn First People's Hospital, HuaiAn, Jiangsu
  - WuXi People's Hospital, Wuxi, Jiangsu

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Vose J, Armitage J, Weisenburger D; International T-Cell Lymphoma Project. International peripheral T-cell and natural killer/T-cell lymphoma study: pathology findings and clinical outcomes. J Clin Oncol. 2008 Sep 1;26(25):4124-30. doi: 10.1200/JCO.2008.16.4558. Epub 2008 Jul 14. PMID 18626005
- [Background] Coleman M, Martin P, Ruan J, Furman R, Niesvizky R, Elstrom R, George P, Kaufman TP, Leonard JP. Prednisone, etoposide, procarbazine, and cyclophosphamide (PEP-C) oral combination chemotherapy regimen for recurring/refractory lymphoma: low-dose metronomic, multidrug therapy. Cancer. 2008 May 15;112(10):2228-32. doi: 10.1002/cncr.23422. PMID 18338745
- [Background] Ning ZQ, Li ZB, Newman MJ, Shan S, Wang XH, Pan DS, Zhang J, Dong M, Du X, Lu XP. Chidamide (CS055/HBI-8000): a new histone deacetylase inhibitor of the benzamide class with antitumor activity and the ability to enhance immune cell-mediated tumor cell cytotoxicity. Cancer Chemother Pharmacol. 2012 Apr;69(4):901-9. doi: 10.1007/s00280-011-1766-x. Epub 2011 Nov 12. PMID 22080169
- [Background] Shi Y, Dong M, Hong X, Zhang W, Feng J, Zhu J, Yu L, Ke X, Huang H, Shen Z, Fan Y, Li W, Zhao X, Qi J, Huang H, Zhou D, Ning Z, Lu X. Results from a multicenter, open-label, pivotal phase II study of chidamide in relapsed or refractory peripheral T-cell lymphoma. Ann Oncol. 2015 Aug;26(8):1766-71. doi: 10.1093/annonc/mdv237. Epub 2015 Jun 23. PMID 26105599
- [Background] Gong K, Xie J, Yi H, Li W. CS055 (Chidamide/HBI-8000), a novel histone deacetylase inhibitor, induces G1 arrest, ROS-dependent apoptosis and differentiation in human leukaemia cells. Biochem J. 2012 May 1;443(3):735-46. doi: 10.1042/BJ20111685. PMID 22339555
- [Derived] Liang J, Wang L, Wang X, Cui G, Zhou J, Xing T, Du K, Xu J, Wang L, Liang R, Chen B, Cheng J, Shen H, Li J, Xu W. Chidamide plus prednisone, cyclophosphamide, and thalidomide for relapsed or refractory peripheral T-cell lymphoma: A multicenter phase II trial. Chin Med J (Engl). 2024 Jul 5;137(13):1576-1582. doi: 10.1097/CM9.0000000000002836. Epub 2023 Dec 10. PMID 37839894